CLINICAL TRIAL: NCT04086355
Title: Effect of Masticatory Electrical Stimulation on Dysphagia in Spastic Cerebral Palsy
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, amira farag, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001630; P.T.REC/012/001630 (Registry Identifier: Research Ehical committee of faculty of pysical therapy); NCT04086355 (Registry Identifier: Clinical Trials.gov Identifier)
Record Dates: First submitted 2019-08-28; First posted 2019-09-11 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Dysphagia
Keywords: Dysphagia; electrical stimulation; cerebral palsy
MeSH Terms: conditions — Deglutition Disorders; Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: two parallel groups ,study group received oro motor exercise and neuromuscular electrical stimulation on masseter and digastric muscles.control group received the same but placebo electrical stimulation.
Who Masked: Participant
Masking Description: participants did not have knowldge if they in study or in control group ,as the exercises applied the same in both group and electrical stimulation the same ,the device turn on in both groups but their is no real signals reached to control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of electrical stimulation on dysphagia in cp (Experimental): the study group that was treated by selected oromotor exercise program in addition to neuromuscular electrical stimulation, Feeding level progress was evaluated by functional oral intake scale,oro motor skills were evaluate by oromotor assessment scale, weight gain and height were measured pre and post 2 months of the treatment.
  Interventions: Other: oromotor exercises and neuromuscular electrical stimulations
- effect of oromotor exercise on dysphagia in cp (Experimental): the control group was treated by the same oromotor exercise program in addition to placebo effect of neuromuscular electrical stimulation. Feeding level progress was evaluated by functional oral intake scale,oro motor skills were evaluate by oromotor assessment scale, weight gain and height were measured pre and post 2 months of the treatment.
  Interventions: Other: oromotor exercises and neuromuscular electrical stimulations

INTERVENTIONS:
Other: oromotor exercises and neuromuscular electrical stimulations — treatment study group with occupational exercises and electrical stimulation
  Other Names: occupational therapy and physical agents

SUMMARY:
This study was conducted to evaluate the effectiveness of masticatory muscles electrical stimulation on oromotor skills, feeding level progress and child growth in children with dyaphagia. Forty children diagnosed as spastic cerebral palsy, from both genders, age ranging from 2 to 5 years were enrolled in the current study. They were randomly allocated in to study group (A) received oromotor exercises and neuromuscular electrical stimulation on masseter and digastric muscles and control group (B) received same exercises but placebo electrical stimulation. The result showed significant improvement in all variables in both groups. However, the study group showed significant different in feeding level in compare with control group.

DETAILED DESCRIPTION:
Study design:

A randomized controlled clinical trial was conducted after interviews were done with the parents or care givers of all children, before starting the study to demonstrate the aim, procedures and potential benefits of the study. Children' parents provided written informed consent before the study was conducted.

Participants:

Forty spastic CP children (26 girls and 14 boys), age ranging from 2 to 5 years, participated in this study. They were selected based on the following criteria; having at least score (level 4) according to functional oral intake scale (FOIS), and they had good head control. Children were excluded if they had; oral hypersensitivity, acute or chronic dental problems, released primitive reflexes as asymmetrical tonic neck reflex or Seizures.

Participants who met the eligible criteria were assigned randomly to either study or control group of equal numbers. Each child in both groups received an oro-motor exercises program as home routine 3 times daily before each meal. Children in the study group received 20-minutes of neuromuscular electrical stimulation (NMES) (multi current SND 64227) which consisted of two-channels electrotherapy system designed for neuromuscular rehabilitation. The NMES was applied with 60 Hz of 230 milliseconds twice weekly for 8 weeks. While participants in the control group received placebo NMES.

Procedures:

Assessment:

1. weight and height Weight and height of each child were measured pre and post treatment by using weight and height measuring scale.
2. Feeding level Dysphagia feeding level was assessed by using functional oral intake scale (FOIS) , taking into consideration that tube dependent children at levels from 1-3 were excluded from the study).
3. Assessment of oromotor skills by oromotor assessment scale (OMAS).

Treatment:

Home routine exercises The exercises were demonstrated to the parents to warrant the uniformity of the training program. They were instructed to conduct the exercises three times daily before each meal. This home routine included passive movement, active movement and sensory stimulation.

1. Passive movement exercises:

   Passive movement included massage and passive range of motion (ROM) exercises. A-Massage: for gums, cheeks, lips and tongue for ten repetitions.
   * Gum massage: upper and lower gum massage started from middle of the gum to the end in the right and left side using regular brush.
   * Lip massage: started from side to side, it was applied for the upper then the lower lips.
   * Cheek massage: Applied intra oral in a circular way.
   * Tongue massage: Applied in the lateral side of the tongue from backward to forward direction in the right and left side using regular tooth brush.

   B-Passive range of motion was done for jaw, tongue and lips for ten repetitions.
   * Jaw movement: cupping lower jaw and move it up and down.
   * Tongue movement: Moving tongue laterally (right and left) and upward directions were done by tongue depressor and fingers.
   * Movement for lip closure: pushing the lips passively against each other like a kissing position.
2. Active movements:

   Active movement included active ROM for jaw, cheeks and lips and stretching for lips.

   A-Active ROM
   * Active jaw ROM: Jaw closure against resistance through biting on tongue depressor and holding for 6 seconds with ten times repetition.
   * Active cheek ROM: Cheek compress by drinking from straws with different diameters.

   B- lip stretching; Stretching upper and lower lips sustain twenty seconds for three sets.
3. Sensory stimulation; Sensory stimulation was done through Lollipop exercise by stimulation of lip closure, cheek and tongue movement through moving the lollipop in different directions.

Neuromuscular electrical stimulation The NMES was applied by the neo-faradic stimulation (Two channels system. The electrodes were applied bilaterally. The first channel was applied over the neck between the hyoid and jaw, (approximately on the belly of the digastric muscle). The second channel was applied on the side of the face, (approximately on the masseter muscle). The intensity level was determined by visible muscle contractions without pain sensation. For children in the study group, the intensity level was from 7 mA to 15 mA, the time of rise and fall was equal (50% raise and 50% fall) and the time on and off was fixed as; 3,1s:3,1s. While those in the control group received placebo NMES without any signals reached to the muscles.

All children received the treatment sessions 20 minutes, twice/weekly for 2 months in addition to home routine exercises.

Statistics:

Paired and unpaired t-test were conducted for comparison of the mean and slandered deviation for the demographic characteristics, weight gain and height variables. Mann-Whitney U test was conducted for comparison of median values of FOIS between both groups. Wilcoxon Signed Ranks Test was conducted for comparison between pre and post treatment median values of FOIS in each group.

The level of significance for all statistical tests was set at p < 0.05. All statistical measures were performed through the statistical package for social studies (SPSS) version 22 for windows.

Results:

General characteristics of participants:

The pretreatment comparison between both groups showed insignificant difference regarding the mean values of age, weight and height (p<0.05).

Regarding weight gain and height there was insignificant difference between both groups before and after treatment (p>0.05). While pre and post treatment within group comparison revealed significant difference in both groups (p<0.05).

Regarding the feeding level (FOIS) comparison of values between both groups considering the feeding level showed a statistically significant difference in each group after treatment. While between both groups, there was insignificant difference before treatment (p>0.05). After treatment, there was significant difference between the study and the control groups in FOIS (p<0.05).

Regarding to oromotor skills There was insignificant difference between both groups before and after treatment (p>0.05), While a significant different was in each group after treatment when comparing it with its pretreatment value was recorded (p<0.05)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic cerebral palsy.
* age ranged from 2 to 5 years.
* They had score level 4 or more according to functional oral intake scale (FOIS)
* They had head control

Exclusion Criteria:

* oral hypersensitivity.
* any acute or chronic dental problems
* released primitive reflexes as asymmetrical tonic neck reflex.
* seizures
* genetic syndrome

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
feeding level progress | time of treatment was two months
  functional feeding level evaluated with functional oral intake scale .this scale contain one item (feeding level) .the score ranging from level one to level seven seven levels ,the best level is level seven ( total oral intake without restrictions) the worth level is level one 9tube dependent .the final score is the number of level .assessed pre and post treatment
oromotor skills | period of treatment was two months
  oro motor assessment scale assess oromotor skills , it has seven items each item has four scores from zero to three, zero the worth and three the best. Each item was assessed 30 s. Their was no interfering with the way the caregiver or the child ingested the food, When the child presented more than one type of oral motor skill for the same item, the most frequently used skill was considered during the assessment. The final classification score of oral motor skill was attributed based on the most frequent score and if there was a tie between two scores, the highest score determined the diagnosis of the predominant type oro motor skills assessed pre and post ttt
weight gain | period of treatment was two months
  assess weight pre and post ttt by weight measuring scale.Child who able to stand was asked to stand on the weight measuring scale and record the weight of the child as show in The child who unable to stand assess weight of mother while carrying the child and record the weight then assess weight of mother alone and record her weight also ,then substract to find the weight of child in kg
height | period of treatment was two months
  assess height pre and post ttt by height measuring scale.Child who able to stand was asked to stand on the height measuring scale and elevate the arm of the height measuring scale till the vertex of the child then the height was recorded. child who unable to stand ask mother to lie the child supine line position then take land mark from the far point of the head , then take also land mark from the most far point from the heel and keep knee extended, after that measure the distance between two land mark and record the height in cm .

CONTACTS AND LOCATIONS:
Locations (1):
- Out Patient Clinic Faculty of Physical Therapy Cairo University, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.